CLINICAL TRIAL: NCT01075789
Title: The Combined Use of Intranasal Lignocaine Spray and Oral Lignocaine Gel to Reduce the Pain and Trauma Associated With Nasogastric Tube Insertion in Hospitalised Children.
Brief Title: Using Lignocaine Spray and Gel to Reduce the Pain Associated With Nasogastric Tube Insertion in Children
Acronym: NGTIPPS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: The University of Queensland (Other)
Responsible Party: Principal Investigator, Dr Stephen Lambert, Senior Research Fellow, The University of Queensland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NGTIPPS
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Intubation; Difficult
Keywords: Pain; Discomfort; Insertion; Nasogastric tube
MeSH Terms: conditions — Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): This arm will include children aged 6 years of age and older seen at the Royal Children's Hospital who are having an NGT inserted for a clinical indication and who have never experienced an NGT insertion before. These children will be randomised to be in this placebo arm or the treatment arm in a 1:1 ratio. The placebo for swallowing is a viscous, coloured, sucrose-flavoured gel designed to match the appearance of the treatment lignocaine gel to be swallowed by the treatment arm, and normal saline will be delivered to the nasal turbinates and nasopharynx in a similar way to atomised xylocaine in the treatment arm.
  Interventions: Drug: Placebo
- Lignocaine (Active Comparator): This arm will include children aged 6 years of age and older seen at the Royal Children's Hospital who are having an NGT inserted for a clinical indication and who have never experienced an NGT insertion before. These children will be randomised to be in this treatment placebo arm or the treatment arm in a 1:1 ratio. The children in the treatment arm will receive xylocaine viscous 2% to swallow, and atomised 10% xylocaine to the nasal turbinates and nasopharynx.
  Interventions: Drug: Lignocaine
- Pre/post intervention evaluation group (Active Comparator): This is a contemporaneous arm of children aged 6 years of age and older requiring nasogastric intubation for a clinical reason, who have previously had a nasogastric tube inserted. These children will be ask to rate by recall their previous NGT intubation on a VAS pain scale, and then will perform a post-procedure VAS pain assessment.
  Interventions: Drug: Lignocaine

INTERVENTIONS:
Drug: Lignocaine — Lignocaine 10% solution administered intra nasally plus lignocaine 2% solution administered orally.
  Arms: Lignocaine; Pre/post intervention evaluation group
Drug: Placebo — Viscous, coloured, sucrose flavoured gel solution to match xylocaine viscous in appearance, normal saline administered intranasally to the nasal turbinates and nasopharynx.
  Arms: Placebo

SUMMARY:
Nasogastric tube insertion is one of the most common invasive procedures performed in children's hospitals, and has long been recognised as one of the most traumatic and painful. As a once off procedure, a nasogastric tube insertion is extremely distressing but the repeated procedures that many children endure as a necessary part of treatment for a chronic disease can be so traumatic that psychological damage may occur. There have been a limited number of studies carried out which have looked at methods to reduce the pain and trauma associated with this procedure, but most of these have been carried out in the adult population.

The investigators propose to carry out a research project in a paediatric setting to definitively investigate the use of local anaesthetic spray, in combination with local anaesthetic gel, to numb the nasal passages and the back of the throat, with the aim of reducing or removing the unpleasant sensation of the nasogastric tube placement. If the study shows a benefit from the use of local anaesthetics, it would be an inexpensive and easily incorporated intervention that could be inserted into the routine procedure for nasogastric tube insertion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parent of guardian
2. Signed assent from subject
3. Subject must have insertion of a nasogastric tube ordered as part of his/her current treatment
4. Must be 6 years of age or older
5. Must be able to complete visual analogue scale (VAS)

Exclusion Criteria:

1. Congenital abnormalities of the naso/oropharyngeal area
2. Any surgical alterations in the naso/oropharyngeal area
3. Mucositis
4. Known history of hypersensitivity to xylocaine or other local anaesthetics
5. Known history of hypersensitivity to other components of the xylocaine solutions such as methyl or propyl hydroxybenzoate, ethanol, polyethylene glycol 400, banana flavour PHL-131980, menthol, saccharin
6. Allergy to food colouring
7. Presence of tracheotomy / tracheostomy
8. Presence of tumour in the nasopharyngeal/oropharyngeal area
9. Impaired gag reflex
10. Impaired swallow
11. Any cardiac condition
12. Diabetes
13. Hypertension
14. Current use of antidepressant medication
15. Current use of cimetidine or propranolol
16. Significantly impaired liver function
17. Significantly impaired renal function
18. Current use of anti-arrhythmic medication

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Reduction in mean visual analogue scores (VAS) in study arm | 10 minutes following nasogastric tube intubation

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas T O Neill, BN, Principal Investigator — Royal Children's Hospital, Queensland Paediatric Infectious Diseases Laboratory
Locations (1):
- Queensland Children's Medical Research Institute, Brisbane, Queensland, Australia